CLINICAL TRIAL: NCT00836810
Title: Circadian Variation in Cytokines and the Effect of Timed Release Tablet Prednisone in Polymyalgia Rheumatica
Brief Title: Timed Release Tablet Prednisone in Polymyalgia Rheumatica
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME/2008/3031
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Polymyalgia Rheumatica
Keywords: Circadian variations of cytokines in PMR; effect of TRT Prednisone in cytokines
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timed Release Tablet Prednisone (Experimental): 12 patients will be taking the intervention night time timed release tablet (TRT) prednisone at a dose of 7mg a day over 2 weeks.
  Interventions: Drug: Timed Release Tablet Prednisone
- Standard Prednisolone (Active Comparator): 12 patients will be taking morning Prednisolone at a dose of 7mg over 2 weeks.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Timed Release Tablet Prednisone — Dose: 7mg, taken at 10pm every night for 2 weeks in the form of oral tablets.
  Other Names: Lodotra
  Arms: Timed Release Tablet Prednisone
Drug: Prednisolone — Dose: 7mg, taken in the morning for 2 weeks in the form of oral tablets.
  Arms: Standard Prednisolone

SUMMARY:
Polymyalgia Rheumatica (PMR) is a disease that usually affects older people. Patients complain of stiffness and pain around the shoulders and hips. The stiffness is more severe in the morning.

Research in Rheumatoid Arthritis (RA), which is also much worse in the mornings, has shown that IL-6 (a chemical messenger) peaks in the morning with very low levels in the evening. This may explain why stiffness is most severe in the morning. The investigators have recently shown that timed release tablet (TRT) prednisone reduced morning IL-6 levels close to normal in RA patients.

In PMR, IL-6 levels are high. Given that both RA and PMR have the same variation of symptoms (worse in the morning); it's likely that PMR patients have the same variation in IL-6 levels. In a pilot study of 4 patients conducted within our department, IL-6 levels did, indeed, show a pattern similar to that found in RA patients, but the number of patients is small and the results need to be confirmed.

PMR is treated with moderate doses of glucocorticoid for about 2 years. While generally abolishing symptoms, these doses are very likely to cause adverse effects such as high blood pressure, weight gain and diabetes. These side effects are much less frequent when lower doses are used but these are not sufficient to control PMR using traditional dosing regimes.

Therefore, the investigators wish to investigate whether TRT prednisone in PMR will reduce IL-6 and morning symptoms similar to those in RA. The investigators think that it will do so, and will achieve symptomatic relief at a lower dose. If this is the case, then treating patients with lower doses may mean reduced risk of glucocorticoid induced side effects in the future.

Patients will be recruited through the outpatient clinics at the University Hospitals Bristol, NHS Foundation Trust, Rheumatology Centre. Each patient will give fully informed consent after being given details of the study and a patient information sheet. The research doctor will take the consent 2-5 days after this information has been provided and with the presence of a witness. The study will consist of the collection and analysis of sequential blood samples over a 24 hour period on 2 occasions 2 weeks apart, taking TRT prednisone 7 mg / standard release prednisolone 7 mg for the intervening period. The investigators will aim to recruit 12 patients in each arm. A single blood sample will be taken when the patient comes for a routine review 2 weeks later.

DETAILED DESCRIPTION:
The volunteers will stay overnight in the Rheumatology Centre; 24-hour Research Facility on two occasions (Night A and Night B) 12-16 days apart. This slight flexibility will allow some leeway in arranging residency nights. In general the investigators will aim for 14 days. After Night A, each volunteer will be randomized (in pre-prepared sealed envelopes) to take one tablet morning or evening. Half the patients will take active standard release prednisolone in the morning. The other half will receive active TRT Prednisone 7mg to be taken each evening at 22:00 until the day after Night B. All study medication will then be discontinued and standard therapy (prednisolone 15mg each morning) commenced. Patients will be reviewed after 2 weeks to ensure expected clinical response and to measure IL-6 and other cytokines in the blood sample that is also needed to check the acute phase response.

On Night A and Night B, volunteers will attend the Rheumatology Centre at 15:00.

First, standard assessment tools will be used by the research doctor to assess the state of the patient's condition.

These assessments will be:

* Morning stiffness (minutes)
* Pain (visual analogue scale)
* Patient's opinion of condition
* Clinician's opinion of condition
* Health Assessment Questionnaire
* BRAF-MDQ fatigue scale and the Hospital Anxiety and Depression Scale.

An intravenous (IV) cannula will be inserted into the elbow area. At least one hour after the IV cannula is placed, but usually at 16:30, a blood sample (2ml) will be taken through the IV cannula and the cannula flushed. At 22:30 the main lights will be switched off and the volunteer encouraged to sleep. In total, 20 samples will be taken from the cannula over 24 hours.

The investigators will calculate mean and standard deviation (or non-parametric analysis if the data are not normally distributed) for blood cytokines for each time point. These mean and standard deviations will be compared for pre- and post-TRT prednisone samples.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMR by standard criteria. The Bird criteria will be used. 3 or more features are required to make the diagnosis.

  * Bilateral shoulder pain/stiffness
  * Duration of symptoms <2/52
  * Initial ESR >40 mm/h
  * Stiffness >1 h
  * Age >65 years
  * Depression and/or weight loss
  * Bilateral upper arm tenderness
* Are over 50 but less than 85 years old.
* No or stable NSAID or analgesic therapy for at least 7 days.
* Currently active disease defined by a CRP at least 10mg/L, ESR at least 29mm in one hour or PV >1.72

Exclusion Criteria:

* Currently on oral glucocorticoid treatment or taken within 2 months
* Parenteral glucocorticoid treatment with the last 2 months
* Pregnancy and lactation
* Inflammatory diseases such as inflammatory bowel disease, colitis, asthma
* Co-existent giant cell arteritis
* Other auto-immune diseases
* Cancer
* Infections, treatment with antibiotics within the past 6 weeks
* Significant renal disease (creatinine >150 μmol/L)
* Significant hepatic impairment
* Participation in a clinical trial within the past 30 days
* Working shift employee
* Jet lag

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Kirwan, MBBS,MD,FRCP, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (1):
- University Hospitals Bristol NHS Trust, Bristol, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 35 sequential eligible patients invited to participate 12 agreed to do so.
Pre-assignment Details: One patient was a technical failure (unable to take 24 hour blood samples) before the treatment randomisation step, leaving 11 patients included.
Groups:
- Timed Release Tablet Prednisone: 11 patients will be taking the intervention night time timed release tablet (TRT) prednisone at a dose of 7mg a day over 2 weeks.
  Timed Release Tablet Prednisone: Dose: 7mg, taken at 10pm every night for 2 weeks in the form of oral tablets.
- Standard Prednisolone: 11 patients will be taking morning Prednisolone at a dose of 7mg over 2 weeks.
  Prednisolone: Dose: 7mg, taken in the morning for 2 weeks in the form of oral tablets.
Period: Overall Study
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Started | 5 | 6
Completed | 4 (1 patient was subsequently diagnosed with SLE and, per protocol, was not included.) | 6
Not Completed | 1 | 0
Not completed — New diagnosis | 1 | 0

BASELINE CHARACTERISTICS:
Population: Fewer participants were recruited than anticipateed within the time frame of the trial.
Groups:
- Timed Release Tablet Prednisone: Patients will be taking the intervention night time timed release tablet (TRT) prednisone at a dose of 7mg a day over 2 weeks.
  Timed Release Tablet Prednisone: Dose: 7mg, taken at 10pm every night for 2 weeks in the form of oral tablets.
- Standard Prednisolone: Patients will be taking morning Prednisolone at a dose of 7mg over 2 weeks.
  Prednisolone: Dose: 7mg, taken in the morning for 2 weeks in the form of oral tablets.
- Total: Total of all reporting groups
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Median (Full Range); unit: years] | 77.5 [67 to 79] | 72.5 [67 to 79] | 76 [67 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 6 | 10
plasma IL-6 peak values (pg/ml) [Mean (Standard Deviation); unit: pg/ml] | 53.5 (46.7) | 40.1 (22.3) | 45.5 (32.4)
plasma IL-6 AUC [Mean (Standard Deviation); unit: pg*hr/ml] | 191 (232) | 236 (246) | 218 (228)
plasma viscosity (mPa.s) [Median (Full Range); unit: mPa.s] | 1.77 [1.73 to 1.9] | 1.875 [1.75 to 2.13] | 1.8 [1.73 to 2.13]
Morning stiffness [Mean (Standard Deviation); unit: minutes] | 75 (38.7) | 115 (55) | 96.7 (48.3)
Pain [Mean (Standard Deviation); unit: mm] — VAS 0mm (better) -100mm (worse)
  mm | 54.8 (23.6) | 62.2 (15.0) | 59.2 (25.1)
Patient's opinion of condition [Mean (Standard Deviation); unit: VAS 0mm (better) - 100mm (worse)] | 54.8 (29.3) | 64.2 (16.3) | 60.4 (21.4)
Clinician's opinion of disease activity [Mean (Standard Deviation); unit: VAS 0mm (better) - 100mm (worse)] | 54.8 (23.6) | 62.0 (15.0) | 59.1 (18.0)
Polymyalgia Rheumatica Disease Activity Score [Mean (Standard Deviation); unit: units on a scale] — PMR Disease Activity Score (PMR-AS). Formula:
  PMR-AS = C-reactive protein (mg/L) + visual analogue scale, patient (0[better]-10[worse] cm) + visual analogue scale, physician (0[better]-10[worse] cm) + morning stiffness (min) x 0.1 + elevation of the upper limbs (3 = none; 2 = below shoulder girdle; 1 = up to shoulder girdle; 0 = above shoulder girdle)
  A score below 7 implies low disease activity, a score range of 7 - 17 reflects medium activity and a score of more than 17 indicates an active disease.
  units on a scale | 29.1 (8.7) | 47.1 (22.2) | 39.9 (19.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Serum IL-6 Concentration
Description: Pre-treatment (Night A) peak minus post-treatment (Night B) peak. Peaks defined as the highest value for each patient from measures at 0, 1.5, 3, 4.5, 5.5, 6.5, 7.5, 8.5, 9.5, 10.5, 11.5, 12.5, 13.5, 14.5, 15.5, 17, 19, 20.5, 22, and 24 hours after 16.30 on day before treatment (Night A) and last day of treatment (Night B) and the peak identified for each one.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Number analyzed (Participants) | 4 | 6
pg/ml | 11.5 (8.3) | 29.3 (15.1)
Statistical Analysis 1: Comparison: Timed Release Tablet Prednisone; Test type: Superiority; p < 0.001, t-test, 2 sided — A priory test for statistical significance was P<0.05
Statistical Analysis 2: Comparison: Standard Prednisolone; Test type: Superiority; p < 0.001, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 3: Comparison: Timed Release Tablet Prednisone vs Standard Prednisolone; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — A priori statistical significance set as P<0.05

2. Primary Outcome: Change in Area Under the Curve (AUC) of Plasma IL-6
Description: Pre-treatment (Night A) AUC minus post-treatment (Night B) AUC. AUC calculated from measures at 0, 1.5, 3, 4.5, 5.5, 6.5, 7.5, 8.5, 9.5, 10.5, 11.5, 12.5, 13.5, 14.5, 15.5, 17, 19, 20.5, 22, and 24 hours after 16.30 on day before treatment (Night A) and last day of treatment (Night B).
Time Frame: 24 hour measurements 2 weeks apart
Measure: Mean (Standard Deviation); unit: pg*hr/ml
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Number analyzed (Participants) | 4 | 6
pg*hr/ml | 113.5 (77.7) | 97.9 (84.3)
Statistical Analysis 1: Comparison: Timed Release Tablet Prednisone; Test type: Superiority; p < 0.001, t-test, 2 sided; A priori statistical significance set at P<0.05
Statistical Analysis 2: Comparison: Standard Prednisolone; Test type: Superiority; p < 0.01, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 3: Comparison: Timed Release Tablet Prednisone vs Standard Prednisolone; Test type: Superiority; p < 0.01, t-test, 2 sided — A priori statistical significance set at P<0.05

3. Secondary Outcome: Percentage Change in Morning Stiffness
Description: How long was your morning stiffness today? Pre-treatment (Night A) value minus post-treatment (Night B) value divided by pre-treatment value.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline morning stiffness
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Number analyzed (Participants) | 4 | 6
percentage of baseline morning stiffness | 75.0 (38.7) | 115.0 (55.0)
Statistical Analysis 1: Comparison: Timed Release Tablet Prednisone; Test type: Superiority or Other; p = 0.023, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 2: Comparison: Standard Prednisolone; Test type: Superiority; p = 0.0906, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 3: Comparison: Timed Release Tablet Prednisone vs Standard Prednisolone; Test type: Superiority; p = 0.044, t-test, 2 sided — A priori statistical significance set at P<0.05

4. Secondary Outcome: Pain (Severity)
Description: 100mm visual analogue scale. Question: How much pain have you had in the last 24 hours? Anchors: No pain; Severe pain. Min score 0, Max score 100. Higher value is worse outcome.
Time Frame: 24 hour period after 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Number analyzed (Participants) | 4 | 6
mm | 26.5 (25.3) | 19.5 (13.1)
Statistical Analysis 1: Comparison: Timed Release Tablet Prednisone; Test type: Superiority; p = 0.007, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 2: Comparison: Standard Prednisolone; Test type: Superiority; p = 0.002, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 3: Comparison: Timed Release Tablet Prednisone vs Standard Prednisolone; Test type: Superiority; p = 0.57, t-test, 2 sided — A priori statistical significance set at P<0.05

5. Secondary Outcome: Patient's Opinion of Condition
Description: 100mm visual analogue scale. Question: Considering all the ways your pain and/or stiffness affect(s) you, please mark on the line how well you are doing. Anchors: Very well; Very badly. Min 0 Max 100 (poor outcome).
Time Frame: Current value at baseline and after 2 weeks treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Number analyzed (Participants) | 4 | 6
mm | 17.8 (20.6) | 26.0 (17.6)
Statistical Analysis 1: Comparison: Timed Release Tablet Prednisone; Test type: Superiority; p = 0.022, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 2: Comparison: Standard Prednisolone; Test type: Superiority; p = 0.002, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 3: Comparison: Timed Release Tablet Prednisone vs Standard Prednisolone; Test type: Superiority; p = 0.51, t-test, 2 sided — A priori statistical significance set at P<0.05

6. Secondary Outcome: Clinician's Opinion of Disease Activity.
Description: 100mm visual analogue scale. Question: Clinician's opinion of disease activity. Anchors: None; Severe Min 0 Max 100 (worse)
Time Frame: Current at baseline and after 2 weeks treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
Number analyzed (Participants) | 4 | 6
mm | 19.0 (18.1) | 20.3 (9.3)
Statistical Analysis 1: Comparison: Timed Release Tablet Prednisone; Test type: Superiority; p = .003, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 2: Comparison: Standard Prednisolone; Test type: Superiority; p = .001, t-test, 2 sided — A priori statistical significance set at P<0.05
Statistical Analysis 3: Comparison: Timed Release Tablet Prednisone vs Standard Prednisolone; Test type: Superiority; p = 0.88, t-test, 2 sided — A priori statistical significance set at P<0.05

ADVERSE EVENTS:
Time Frame: 2 week duration of treatment and 2 weeks of standard treatment.
Arm/Group | Timed Release Tablet Prednisone | Standard Prednisolone
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Small number of patients not blind to study treatment which may have influenced reports of morning stiffness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No